CLINICAL TRIAL: NCT03882307
Title: Association of Serum Interleukin -6 and Transforming Growth Factor Beta Levels With Response to Antiviral Therapy for Chronic Hepatitis c Patients
Brief Title: Levels of Interleukin-6 andTransforming Growth Factor Beta in HCV Patients Sera
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hayam Hamdy Mahmoud, principle investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: hhayam
Record Dates: First submitted 2019-03-15; First posted 2019-03-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C virus therapy; interleukin-6; transforming growth factor -beta; sustained virological response
MeSH Terms: conditions — Hepatitis C, Chronic; Camurati-Engelmann Syndrome | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Intervention Model Description: assess serum level of interleukin-6 and transforming growth factor beta before intervention and after intervention with sofosbuvir and daclatasvir.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- group1 (naive) (No Intervention): Assess serum level of interleukin-6 and transforming growth factor beta before the course of treatment
- group2 (sustained responder) (Active Comparator): Assess serum level of interleukin-6 and transforming growth factor beta after three months from the end of treatment Sofosbuvir (SOF) (400 mg once per day) and daclatasvir (DCV)(60mg once per day) or simeprevir (SIM) (150 mg once per day) for 3 months treatment regimens
  Interventions: Drug: sofosbuvir and daclatasvir

INTERVENTIONS:
Drug: sofosbuvir and daclatasvir — oral tablets
  Other Names: Sovaldi
  Arms: group2 (sustained responder)

SUMMARY:
Hepatitis C virus (HCV) infection is associated with significant morbidity and mortality owing to progression of a high percentage (85%) of HCV infected patients to chronic hepatitis, which might lead to the development of liver cirrhosis or hepato cellular carcinoma..

Egypt has possibly the highest HCV prevalence in the world, 10-20% of the general population .

DETAILED DESCRIPTION:
Currently, second-generation direct-acting antiviral agents have been used for chronic hepatitis C treatment. The association of sofosbuvir with daclatasvir or simeprevir , with or without ribavirin , directly inhibits viral replication .

Sofosbuvir (400 mg once per day) and daclatasvir (60mg once per day) or simeprevir (150 mg once per day) for 3 months treatment regimens.

Sofosbuvir-based antiviral therapy guarantees efficacy in HCV eradication in approximately 90% of cases and is associated with mild to moderate adverse effects.

Overall, studies describe an increase in serum cytokine levels in chronic hepatitis C patients, when compared with healthy individuals. ,interleukin-6(IL-6) is produced mainly by kupffer cells and induces the production of the acute phase proteins, C-reactive protein and haptoglobin .

Previous studies reported that serum Interleukin-6 levels were increased, compared with healthy individuals, in patients with some liver diseases.Previous results suggest that baseline levels of Interleukin, as well as their decrease during treatment .Transforming growth factor beta (TGF-β) is a cytokine that has been assigned a key role in epithelial repair. Injury to the liver elicits a rapid increase in its expression. HCV -infected hepatocytes produce (TGF-β) which may stimulate T-regulatory cells.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years.
* HCV RNA positivity .
* Any Body Mass Index(BMI).
* Treatment-naive or treatment experienced.
* all fibrosis stages.

Exclusion criteria:

* Direct serum bilirubin greater than 2 mg/dl.
* Serum albumin less than 2.8 g/dl.
* International normalization ratio (INR) greater than or equal to 1.7
* Platelet count less than 50 000/mm3.
* Ascites or history of ascites.
* Hepatic encephalopathy or history of hepatic encephalopathy.
* Hepatocellular carcinoma.
* Serum creatinine greater than 2.5 mg/dl .
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
mean difference in level of interleukin-6 and transforming growth factor beta after treatment | three months from the end of treatment
  serum level of interleukin-6 and transforming growth factor beta will be measured before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: hayam hamdy, master deree, Principal Investigator — faculty of medicine,medical microbiology department
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Serum concentrations of(IL-6 and TGF-β) will be measured before treatment and after three months from the end of the course of treatment with sofosbuvir 400 mg once daily plus daclatasvir 60 mg for three months using a commercially available Quanti kine ELISA (Enzyme linked Immune sorbent Assay ).

REFERENCES:
- [Background] Rahman El-Zayadi A, Abaza H, Shawky S, Mohamed MK, Selim OE, Badran HM. Prevalence and epidemiological features of hepatocellular carcinoma in Egypt-a single center experience. Hepatol Res. 2001 Feb;19(2):170-179. doi: 10.1016/s1386-6346(00)00105-4. PMID 11164741
- [Background] Sulkowski MS, Gardiner DF, Rodriguez-Torres M, Reddy KR, Hassanein T, Jacobson I, Lawitz E, Lok AS, Hinestrosa F, Thuluvath PJ, Schwartz H, Nelson DR, Everson GT, Eley T, Wind-Rotolo M, Huang SP, Gao M, Hernandez D, McPhee F, Sherman D, Hindes R, Symonds W, Pasquinelli C, Grasela DM; AI444040 Study Group. Daclatasvir plus sofosbuvir for previously treated or untreated chronic HCV infection. N Engl J Med. 2014 Jan 16;370(3):211-21. doi: 10.1056/NEJMoa1306218. PMID 24428467
- [Background] Baskic D, Vukovic VR, Popovic S, Djurdjevic P, Zaric M, Nikolic I, Zelen I, Mitrovic M, Avramovic D, Mijailovic Z. Cytokine profile in chronic hepatitis C: An observation. Cytokine. 2017 Aug;96:185-188. doi: 10.1016/j.cyto.2017.04.008. Epub 2017 Apr 21. PMID 28433893
- [Background] Heinrich PC, Castell JV, Andus T. Interleukin-6 and the acute phase response. Biochem J. 1990 Feb 1;265(3):621-36. doi: 10.1042/bj2650621. No abstract available. PMID 1689567
- [Background] Ueyama M, Nakagawa M, Sakamoto N, Onozuka I, Funaoka Y, Watanabe T, Nitta S, Kiyohashi K, Kitazume A, Murakawa M, Nishimura-Sakurai Y, Sekine-Osajima Y, Itsui Y, Azuma S, Kakinuma S, Watanabe M; Ochanomizu-Liver Conference Study Group. Serum interleukin-6 levels correlate with resistance to treatment of chronic hepatitis C infection with pegylated-interferon-alpha2b plus ribavirin. Antivir Ther. 2011;16(7):1081-91. doi: 10.3851/IMP1864. PMID 22024524
- [Background] Bissell DM, Wang SS, Jarnagin WR, Roll FJ. Cell-specific expression of transforming growth factor-beta in rat liver. Evidence for autocrine regulation of hepatocyte proliferation. J Clin Invest. 1995 Jul;96(1):447-55. doi: 10.1172/JCI118055. PMID 7615817
- [Background] Liaskou E, Wilson DV, Oo YH. Innate immune cells in liver inflammation. Mediators Inflamm. 2012;2012:949157. doi: 10.1155/2012/949157. Epub 2012 Aug 9. PMID 22933833
- See also: related info — https://scholar.google.com/scholar